CLINICAL TRIAL: NCT00153595
Title: A Double-Blind, Randomized Parallel Group, Placebo-Control Study of EW01 in Persistent Allergic Rhinitis (PAR) Patients
Brief Title: EWO1 in Persistent Allergic Rhinitis Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMR93-IRB-90; DOH93-TD-I-1-1-1-006
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2005-09

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Allergic rhinitis; EWO1
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic

INTERVENTIONS:
Drug: EWO1

SUMMARY:
The aim of this double-blind, randomized, parallel group, placebo-controlled study is to assess the efficacy and safety of EWO1 in patients with moderate to severe perennial allergic rhinitis (AR).

DETAILED DESCRIPTION:
Allergic rhinitis is a very common medical problem affecting adults and children alike. It has been estimated that 20% to 25% of the world's population suffer from allergic rhinitis, resulting in considerable morbidity - impaired quality of life. In the U.S., there is an estimated $2.4 billion annual medical cost associated with allergic rhinitis.

In Taiwan, household dust mites (HDM) are primary allergens causing allergic reactions including allergic rhinitis. The incidence of HDM in Taiwan can be as high as 100%. Df, Dp and Blomia tropicalis (Bt) rank among the top 3 most common household dust mites. Antihistamines remain a major therapy for treatment of allergic rhinitis. Chinese herbs have long been used to treat different allergic and immunologic diseases. YU-PING-FENG-SAN (YPFS) with a formulation that contains 3 herbs [Huangqi (HQ), baizhu (BZ), and fangfeng (FF)] has been reported as one of the effective traditional Chinese medicines for the treatment of recurrent rhinitis.

In 3 previous non-placebo controlled clinical studies in perennial rhinitis, it has been demonstrated that by adding Xingyi(XY) to a YPFS formula with CQ, BZ, and FF, additional efficacy benefits can be obtained.

The aim of this double-blind, randomized, parallel group, placebo-controlled study is to assess the efficacy and safety of EWO1 in patients with moderate to severe perennial allergic rhinitis. After a 2-week placebo run-in period, patients who satisfy all of the inclusion/exclusion criteria will be randomized 1:1 to receive either EWO1, or placebo for 28 days. After the treatment-period, patients will be followed for 14 days to see if there is any rebound in rhinitis symptoms. The Primary efficacy endpoint is weekly combined symptom scores at the end of treatment. Besides, intent to treat analyses will be carried out for both efficacy and safety. A minimum of 60 patients will be randomized into this two-treatment parallel-design study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, aged 12 years and above
2. AR confirmed by positive allergen (dust mite; Dp) specific IgE ≧ 2+ within 12 months of enrollment
3. History of persistent moderate to severe allergic rhinitis
4. One or more of the following: abnormal sleep; impairment of daily activities, sports, leisure; problems caused at work or school; and/or troublesome symptoms.
5. Total nasal symptom scores (nasal rhinorrhea, nasal congestion, nasal itching, sneezing and post-nasal drip) ≧ 5 at baseline period (scale 0 : none; 1 : mild; 2 : moderate; 3 : severe)
6. No initiation of immunotherapy within 6 months or no dose change in immunotherapy for 1 month
7. Signed informed consent obtained prior to inclusion into the study

Exclusion Criteria:

1. History of recent (within 6 months) asthma
2. Chronic or intermittent use of inhaled, oral, intramuscular (i.m.), intravenous (i.v.), and/or potent/superpotent topical steroids within 2 weeks
3. Use of prohibited medicines within 2 weeks
4. Use of long-acting antihistamines within 2 weeks
5. Documented evidence of acute or significant chronic sinusitis
6. Chronic use of concomitant medications that could interfere with assessment
7. Known or suspected hypersensitivity to any of the herbal components in EWO1
8. Rhinitis medicamentosa
9. Planned travel outside the study area for a substantial portion of time during the study
10. Use of another investigational product within the past 30 days
11. Pregnant or lactating women; women of child-bearing potential must use adequate contraception.
12. Renal dysfunction as evidenced by creatinine level of 1.5 x upper limit of normal (ULN)
13. Liver dysfunction as evidenced by SGPT of > 1.5 x ULN
14. Signs and symptoms of upper respiratory infection (URI) upon admission

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-11

CONTACTS AND LOCATIONS:
Overall Officials: Min-Chien Yu, Ph.D., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan